CLINICAL TRIAL: NCT05291858
Title: Multidetector Cardiac Computed Tomographic Assessment of Cardiac and Extra Cardiac Vascular Anomalies Associated With Tetralogy of Fallot in Pediatric
Brief Title: Computed Tomographic Assessment of Cardiac and Extra Cardiac Vascular Anomalies Associated With Tetralogy of Fallot
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Rashed Fahmy, assistant lecturer, Assiut University
Other Study IDs: Computed tomography in CHD
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Fallot Tetralogy
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of cardiac and extra cardiac vascular defects associated with Tetralogy of fallot in pediatric patients, regarding frequency and types of anomalies with assesment of multidetector computed tomography diagnostic value.

DETAILED DESCRIPTION:
Tetralogy of Fallot (TOF) is the most common complex cyanotic congenital heart disease (CHD), with a prevalence of 3.5-9%. Almost all pediatric patients born with TOF can now expect to survive to adulthood because of advances in its surgical treatment. In addition to the four diagnostic criteria of TOF that include ventricular septal defect, right ventricular hypertrophy with outflow tract obstruction, and overriding aorta, other extra-cardiac vascular anomalies are frequently coexist . These may involve pulmonary, aortic, and coronary arteries with or without valve abnormalities, aorto-pulmonary vessels, and vena cava connections, is crucial for surgeons in the formulation of surgical strategies. Trans-thoracic echocardiography (TTE) is the initial classical procedure done for these patients, as it can demonstrate heart structure and estimate intra-cardiac pressures, gradients, and contractile functions as well as blood flow direction across any heart defect and emphasizing coronary vessels integrity. However, many extracardiac vascular defects associated with different heart diseases cannot be detected accurately by TTE; consequently, heart catheterization with its invasive complications was widely used for confirming these abnormalities before surgery. Recently, the evolution of multi-slice or multi-detector computed tomography (MDCT) with its multi-planar information, lower doses of radiation, short scanning time, and easy availability suggested it to be a non-invasive reliable diagnostic method for detection of different malformations in pediatric patients with complex CHD. Thus, effective imaging modalities are required to provide a thorough preoperative anatomic description of the associated extracardiac vascular anomalies in pediatric patients with TOF in order to improve surgical planning and outcomes. In recent years, multi-detector computed tomography (MDCT) has become regarded as a reliable non-invasive tool for delineating various anomalies in patients with complex CHD. Few studies have focused on the preoperative evaluation of associated cardiac and extracardiac vascular anomalies in pediatric patients with TOF using MDCT, especially not large case series studies. In this study, we aim to investigate the diagnostic performance of MDCT for assessing associated cardiac and extracardiac vascular abnormalities in patients with TOF.

ELIGIBILITY:
Exclusion criteria

* Non-surgical patients
* Patients with unstable clinical conditions
* Renal insufficiency
* Hypersensitivity to iodinated contrast.

Age range of included patients:

All pediatric patients less than 18 years were included. All patients underwent MDCT and TTE preoperatively. All associated cardiac and extracardiac vascular abnormalities and their percentages will be recorded.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All preoperative TOF patients less than 18 years were included. All patients underwent MDCT and TTE preoperatively. All associated cardiac and extracardiac vascular abnormalities and their percentages will be recorded.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of cardiac and extra cardiac vascular anomalies associated with tetralogy of Fallot by MDCT and its repercussion on preoperative decision. | within a year
  The four main characteristics of TOF [ventricular septal defect, overriding aorta, right ventricular outflow tract (RVOT) obstruction, and right ventricular hypertrophy] and associated cardiac and extracardiac malformations will be analyzed and recorded using a sequential segmental approach. To compare the diagnostic performance of DSCT with that of TTE, we will categorize all the surgically confirmed associated cardiac and extracardiac vascular deformities into five groups, namely abnormal vena cava connection (AVCC), aortic artery and valve disorders, anomalies of the pulmonary artery and valve, deformities of the aortopulmonary vessels, and coronary artery anomalies (CAAs).